CLINICAL TRIAL: NCT06951854
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Therapeutic Exploratory Phase II Clinical Trial to Evaluate the Efficacy and Safety of NV01-A02 in Children With Autism Spectrum Disorder
Brief Title: Phase II Clinical Trial to Evaluate the Efficacy and Safety of NV01-A02 in Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neuroventi Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NV01-A02
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder (ASD
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: NV01-A02 (Experimental): Participants will receive different dose levels of the investigational drug. The drug will be administered orally once daily
  Interventions: Drug: Drug: NV01-A02
- Drug: Placebo (ZP8396) (Placebo Comparator): Participants will receive different dose levels of the investigational drug. The drug will be administered orally once daily
  Interventions: Drug: Drug: Placebo (ZP8396)

INTERVENTIONS:
Drug: Drug: NV01-A02 — NV01-A02 will be administered orally at a different dose once daily for 8 weeks. The formulation is a white, film-coated tablet, designed for use in patients with mild to moderate cognitive impairment.
  Arms: Drug: NV01-A02
Drug: Drug: Placebo (ZP8396) — ZP8396 is a matching placebo tablet administered orally once daily for 8 weeks. The placebo is identical in appearance to NV01-A02 but contains no active ingredient.
  Arms: Drug: Placebo (ZP8396)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, therapeutic exploratory Phase 2 clinical trial designed to evaluate the efficacy and safety of NV01-A02 in pediatric participants diagnosed with Autism Spectrum Disorder (ASD).

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

Children aged 6 to 15 years (inclusive) as of the date of written consent

Individuals who meet all the diagnostic criteria for Autism Spectrum Disorder (ASD) as outlined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)

DSM-5 Diagnostic Criteria for Autism Spectrum Disorder (ASD):

* Persistent deficits in social communication and social interaction across multiple contexts, as manifested by all of the following:

A. Deficits in social-emotional reciprocity

B. Deficits in nonverbal communicative behaviors used for social interaction

C. Deficits in developing, maintaining, and understanding relationships

② Restricted, repetitive patterns of behavior, interests, or activities, as manifested by at least two of the following:

A. Stereotyped or repetitive motor movements, use of objects, or speech

B. Insistence on sameness, inflexible adherence to routines, or ritualized patterns of verbal or nonverbal behavior

C. Highly restricted, fixated interests that are abnormal in intensity or focus

D. Hyper- or hyporeactivity to sensory input or unusual interest in sensory aspects of the environment

③ Symptoms must be present in the early developmental period (but may not become fully manifest until social demands exceed limited capacities, or may be masked by learned strategies later in life)

Exclusion Criteria:

* Individuals weighing less than 16 kg or more than 70 kg

Individuals identified during screening with any of the following medical histories, comorbid conditions, or surgical histories:

* Severe psychiatric disorders (other than autism spectrum disorder) that may affect participation in the clinical trial

  * History of organic brain disease, neurological disorders, or epilepsy/seizures that are not fully controlled by medication or non-pharmacologic surgical treatment (Note: Participants with a history of simple febrile seizures may be included at the investigator's discretion)

    * Severe peripheral arterial disease or coronary insufficiency

      * Presence or history of psychotic symptoms such as delusions or hallucinations (e.g., worsening or recurrence of psychiatric illness)

        * Gastrointestinal diseases (e.g., active peptic ulcers) or history of surgery that may affect absorption of the investigational medicinal product (Note: Participants with a history of simple appendectomy or hernia surgery may be included)

          * Individuals displaying serious self-injurious or aggressive behavior requiring medical intervention during the screening period, as determined by the investigator

            * Individuals with sensory abnormalities such as congenital hearing loss

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the composite scores of the major domains of the Korean Vineland Adaptive Behavior Scales-II (K-Vineland-II) at Week 8 after administration. | From enrollment to the end of treatment at 8 weeks
  Change from baseline in the composite scores of the major domains of the Korean Vineland Adaptive Behavior Scales-II (K-Vineland-II) at Week 8 after administration.*
  For children under 7 years of age, the composite score refers to the standard scores of all four major domains: Communication, Daily Living Skills, Socialization, and Motor Skills.
  For children aged 7 years and older, the composite score refers to the standard scores of the three domains excluding Motor Skills: Communication, Daily Living Skills, and Socialization.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuroventi, Seoul, Seoul, South Korea